CLINICAL TRIAL: NCT06865131
Title: Efficacy Study With StrataXRT for the Prophylaxis of Radiation Dermatitis in Adjuvant Breast Radiation Treatment in Large Breasted Women Using a Prone Technique
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Edward Chow, Co-Principle Investigator with Dr. Irene Karam [ikaram], Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: StrataXRT Prone
Record Dates: First submitted 2024-09-11; First posted 2025-03-07 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Barrier cream; StrataXRT; Prophylaxis; Radiation Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: StrataXRT will be used by the patients daily during their entire treatment, and for a minimum of 2 weeks post-RT. As recommended by the product monograph, patients will be asked to apply StrataXRT twice daily, once in the morning and once in the evening. Additionally, as suggested in the monograph, patients will be directed to reapply the gel any time after they take a shower or if they notice the film is no longer covering the treatment area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- StrataXRT (Experimental): All patients will receive StrataXRT for the duration of their treatment. RT will be delivered as prescribed by the treating radiation oncologist and may include a variety of techniques and beam modifiers. A trained CRA will teach the patient how to apply StrataXRT prior to their first RT at a designated clinic room and will perform daily checks prior to radiation for the first week of treatment to ensure that the patient has covered the entire treatment area. StrataXRT will be used by the patients daily during their entire treatment, and for a minimum of 2 weeks post-RT. As recommended by the product monograph, patients will be asked to apply StrataXRT twice daily, once in the morning and once in the evening. Additionally, as suggested in the monograph, patients will be directed to reapply the gel any time after they take a shower or if they notice the film is no longer covering the treatment area.
  Interventions: Device: StrataXRT

INTERVENTIONS:
Device: StrataXRT — StrataXRT being a silicone-based cream forming a film, it is very flexible and can be applied easily to the prone position and to the contours of the large breast unlike some other barrier film skin interventions

SUMMARY:
For breast cancer patients undergoing adjuvant radiotherapy, radiation dermatitis (RD) is a common occurrence that can negatively impact patients' quality of life (QOL). RD often presents as erythema, pruritus, and/or edema and in more severe cases, skin breakage can occur, resulting in moist desquamation. In a study published it was found that for women with large breasts (n=357), being positioned in the supine position during radiation could lower the rates of moist desquamation from 36.9% in the supine position down to 26.9% when treated in the prone position. Even though the prone position for patients with large breasts did reduce rates of moist desquamation, these results demonstrate that one in five patients still go on to develop severe reactions, even in the prone position. Building on these results, a phase II feasibility study conducted at Sunnybrook, found that the use of a silicone-based film forming topical gel known as StrataXRT could lower the incidence of moist desquamation for patients treated in the prone position even further.

DETAILED DESCRIPTION:
For breast cancer patients undergoing adjuvant radiotherapy, radiation dermatitis (RD) is a common occurrence that can negatively impact patients' quality of life (QOL). RD often presents as erythema, pruritus, and/or edema and in more severe cases, skin breakage can occur, resulting in moist desquamation. In a study published, it was found that for women with large breasts (n=357), being positioned in the supine position during radiation could lower the rates of moist desquamation from 36.9% in the supine position down to 26.9% when treated in the prone position. Even though the prone position for patients with large breasts did reduce rates of moist desquamation, these results demonstrate that one in five patients still go on to develop severe reactions, even in the prone position. Building on these results, a phase II feasibility study conducted at Sunnybrook, found that the use of a silicone-based film forming topical gel known as StrataXRT could lower the incidence of moist desquamation for patients treated in the prone position even further. This currently unpublished study identified that only 10% of patients treated in the prone position using the prophylactic StrataXRT gel experienced grade 2 RD with moist desquamation, and no patients experienced grade 3 RD compared to 26.9% % of patients treated in prone that use the current standard of care moisturizer. Due to StrataXRT being a silicone-based film forming topical gel, it is very flexible and can be applied easily to the prone position and to the contours of the large breast unlike some other barrier film skin interventions.

StrataXRT has previously also been shown to be non-inferior to another silicone-based barrier film known as Mepitel film in the prevention of RD. A study by Chao et al compared the rates of moist desquamation and RD CTCAE scoring in 44 breast cancer patients. Medial and lateral halves of the breast were covered with Mepitel Film and StrataXRT. The results showed no significant differences in the rate of moist desquamation or severity of RD assessed on the CTCAE between groups. This study also noted that nurses had to be responsible for the application of the Mepitel Film, with the average time of application reported to be 15 minutes. In comparison, the StrataXRT was applied and maintained by the patients, and did not require dependency on nursing resources.

Other studies have shown benefits of StrataXRT . A recent randomized control trial published in 2022 by Omidvari et al found that in breast cancer patients (n=100), the use of StrataXRT significantly reduced the mean size of the radiation-induced dermatitis area (p=0.002) when compared to the control group. Additionally, RD as scored by the CTCAE was found to

be significantly more severe in the control group in weeks 1-5, except for week 4 where no significance was indicated. Another randomized control trial (n=49) demonstrated significant differences in the Erythema Index (EI) (p=0.001) and Melanin Index (MI) (p=0.005) between StrataXRT compared to the use of Xderm, a moisturizer. The EI and MI are alternative methods of measuring RD, using electrochemical reflectance most often with a handheld spectrophotometer. However, this tool is not the standard measurement for assessing RD and therefore these results are difficult to compare to other studies. There was no significant difference found between groups using physician assessed outcomes. However, this was likely due to the patient population being at low risk of severe skin reactions, and subsequently no patient in either cohort developed moist desquamation over the course of the study. No added risks or adverse events, other than mild irritation, have been reported following the use of StrataXRT in the aforementioned trials.

In the phase II feasibility study completed at Sunnybrook Odette Cancer Centre, the patient reported outcomes were also favorable and showed promising results for StrataXRT. When analyzing a patient satisfaction questionnaire completed with the prone patients of the study, seven out of eight (88%) patients reported that they felt moderate to high levels of skin protection from StrataXRT. Additionally, all but one patient felt that StrataXRT was easy to apply, and that they had a positive experience with the gel. Patient QOL was evaluated using the Skindex-16 questionnaire, a tool scored out of 96, with a higher score indicating worse QOL overall. In the prone population, the mean total Skindex-16 score was 16.90 out of 96, highlighting that the use StrataXRT was beneficial for patient QoL. In the study conducted by Vesprini et al, secondary outcomes such as clinician-reported grade 2 pain, grade 2 erythema, and grade 1 edema were collected using the CTCAE scale. The incidence of these symptoms was 5.1%, 77.1%, and 48.0% respectively. In the feasibility study on StrataXRT, similar results were extracted using a skin symptom assessment (SSA) and it was found that 10% of patients experienced grade 2 pain, 10% experienced grade 2 erythema, and 10% experienced grade 1 edema. Based on these preliminary results, it is hypothesized that StrataXRT may also lower both erythema and edema substantially.

Due to the limited number of patients in the previous prone cohort (n=10), the investigators would like to consolidate these results by repeating the prone cohort with a larger patient population. The investigators propose to repeat this feasibility study by enrolling 20 additional patients treated in the prone position to confirm these promising results before moving to a phase 3 RCT. Based on the results of our phase II feasibility study, StrataXRT has been well tolerated by patients, is feasible to integrate into daily clinic flow and appears to reduce rates of moist desquamation in patients treated in prone and the incidence of grade 3 radiation dermatitis in this cohort. StrataXRT, though Health Canada approved (License No.: 95612) already, is not commonly used in clinical practice in Canada. There is a need to further study and validate the efficacy of StrataXRT in the prevention of RD for patients with large breasts (minimum of band size of 40 inches or cup size D) treated in the prone position-breast radiation only (boost allowed).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old

  * Informed consent
  * Histological confirmation of breast malignancy (invasive or in situ carcinoma) or phyllodes
  * Patients are scheduled to receive conventionally - (50 Gy/25) or hypofractionated (40 Gy/15) RT to the breast only in the prone position.
  * Women with large breasts equivalent to ≥40-inch band size and/or cup size ≥D
  * Patients treated with or without the addition of boost.
  * Can communicate in English or be aided by a translator

Exclusion Criteria:

* Patients unable to lie prone for the duration of radiation treatment

  * Patient had previous radiation therapy to the treatment area
  * Patients receiving locoregional radiation treatment
  * Patient will receive partial breast external beam radiation or brachytherapy
  * Patients scheduled to receive extreme hypofractionation (26 Gy/5)
  * Patients with active rash, pre-existing dermatitis, or other conditions within the treatment area that may make skin assessment for the study difficult per treating physician discretion.
  * Patients with known allergy or sensitivity to silicone
  * Concomitant cytotoxic chemotherapy
  * Bilateral breast pathology requiring concurrent bilateral breast radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity as defined by the CTCAE V5 assessed by HCP | Once per week during radiation in the treating radiation oncologist's review clinic, and within 3 months following radiation. Radiation treatment duration varies depending on dosage/fractionation, but ranges from 3 to 5 weeks.
  CTCAE Dermatitis Grade:
  0 No symptoms
  1. Faint erythema or dry desquamation
  2. Moderate to brisk erythema; patchy moist desquamation, mostly confined to skin fold and creases; moderate edema
  3. Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion
  4. Life-threatening consequences; skin necrosis or ulceration of full thickness dermis; spontaneous bleeding from involved site; skin graft indicated
  5. Death

SECONDARY OUTCOMES:
Incidence of moist desquamation assessed by HCP | Once per week during radiation in the treating radiation oncologist's review clinic, and within 3 months following radiation. Radiation treatment duration varies depending on dosage/fractionation, but ranges from 3 to 5 weeks.
  Moist desquamation (please circle): No Yes
Radiation-Induced Skin Reaction Assessment Scale (RISRAS) assessed by patient and HCP | Once per week during radiation in the treating radiation oncologist's review clinic, and within 3 months following radiation. Radiation treatment duration varies depending on dosage/fractionation, but ranges from 3 to 5 weeks.
  Researcher component (total score between 0 and 24) Erythema 0(normal skin),1(Dusky Pink), 2(dull red), 3(brilliant red), 4(deep red purple) Dry Desquamation 0(normal skin), 1(<25%), 2(25%-50%), 3 (50%-70%), 4 (>74%) Moist Desquamation 0(normal skin),1.5(<25%), 3.0(25%-50%),4.5 (50%-75%), 6 (>75%) Necrosis 0 (normal skin),2.5(<25%),5.0(25%-50%),7.5(50%-75%),10(>75%) Patient Component Not at all A Little Quite a bit Very much Symptoms Do you have any Tenderness, discomfort 0 1 2 3 or pain of your skin in the treatment area? Does your skin in the 0 1 2 3 treatment area itch? Do you have a burning sensation of your skin 0 1 2 3 in the treatment area? To what extent has your skin reactions and your 0 1 2 3 symptoms affected your day to day activities?
Photographs of treated and non-treated breast/chest wall for blind and unbiased assessment of the skin by HCPs | At baseline when the patient is first recruited, the last treatment day of radiation (3-5 weeks after the first day of radiation depending on radiation dose/fractionation) and at 2 weeks follow up after the end of radiation.
  Photographs of the patient's treated and non-treated breast/chest wall will be taken and used for blind and unbiased assessment of the skin by a group of health care professionals. These results can be compared to in person assessments as scaled on the CTCAE, RISRAS, and the SSA. Patient photos will be taken at baseline when the patient is first recruited, the last treatment day of radiation (3-5 weeks after the first day of radiation depending on radiation dose/fractionation) and at 2 weeks follow up after the end of radiation.
Patient-reported QOL using the Skindex-16 | Once per week during radiation in the treating radiation oncologist's review clinic, and within 3 months following radiation. Radiation treatment duration varies depending on dosage/fractionation, but ranges from 3 to 5 weeks.
  Study ID: ______ Date of assessment (dd/mm/yyyy): ______________ Appointment Type (please circle): baseline last treatment follow-up If follow-up, which follow-up: 2-week 3-month
  During the past week how often Never Bothered Always Bothered have you been bothered by:
  Your skin condition itching 0 1 2 3 4 5 6
  Your Skin condition burning
Patient satisfaction with StrataXRT as assessed by the patient satisfaction questionnaire | During 3 months following radiation
  This survey will consist of negatively and positively phrased questions that will be rated on a four-point Likert scale, in addition to the "not applicable" option.
  Daily activities:
  Please indicate the level of impact StrataXRT has on your ability to ___________: (1=none/no impact, 4= high impact)
  * Perform household chores (laundry, cleaning, cooking, etc.):
    o Not applicable
    1. None
    2. Low
    3. Moderate
    4. High
  * Complete work:
    * Not applicable 1. None 2. Low 3. Moderate 4. High
  * Use transportation (driving, wearing a seatbelt, etc.):
    o Not applicable
    1. None 2. Low 3. Moderate 4. High
  * Exercise:
    o Not applicable
    1. None
    2. Low
    3. Moderate
    4. High
  * Take care of your children, pets, spouse, elderly etc.:
    o Not applicable
    1. None
    2. Low
    3. Moderate
    4. High
  * Sleep:
    o Not applicable
    1. None
    2. Low
    3. Moderate
    4. High
  * Choose clothing to wear:
    o Not applicable
    1. None
    2. Low
    3. Moderate
    4. High
  * Wear a bra:
    * Not applica
Patient-reported skin-related symptoms using the Skin Symptom Assessment (SSA) | Once per week during radiation in the treating radiation oncologist's review clinic, and within 3 months following radiation. Radiation treatment duration varies depending on dosage/fractionation, but ranges from 3 to 5 weeks.
  Study ID: ______ Date of assessment (dd/mm/yyyy): ______________ Appointment Type (please circle): baseline review telephone follow-up If review, what review appointment: 1 2 3 4 5 If telephone follow up, what follow up: 1 2 3 4 5 6 If follow-up, which follow-up: 2-week 3-month Please circle the word that best describes your symptoms in the area receiving radiation right now.
  Pruritus (itchiness) None Mild Moderate Severe Pain or soreness None Mild Moderate Severe Blistering or peeling None Mild Moderate Severe Erythema (redness) None Mild Moderate Severe Pigmentation (discolouration/darkness) None Mild Moderate
HCP reported SSA | Once per week during radiation in the treating radiation oncologist's review clinic, and within 3 months following radiation. Radiation treatment duration varies depending on dosage/fractionation, but ranges from 3 to 5 weeks.
  Study ID: ______ Date of assessment (dd/mm/yyyy): ______________ Completed by: ______________________ Appointment Type (please circle): baseline review follow-up If review, what review appointment: 1 2 3 4 5 If follow-up, which follow-up: 2-week 3-month Photo taken: Y N N/A Please circle the word that best describes symptoms in the area receiving radiation right now.
  Pruritus (itchiness) None Mild Moderate Severe Pain or soreness None Mild Moderate Severe Blistering or peeling None Mild Moderate Severe Erythema (redness) None Mild Moderate Severe Pigmentation (discolouration/darkness) None Mild Moderate Severe Edema (swelling) None

CONTACTS AND LOCATIONS:
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No